CLINICAL TRIAL: NCT00761982
Title: Autologous Bone Marrow Stem Cells in Middle Cerebral Artery Acute Stroke Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Central de Asturias (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OVISEV-01
Record Dates: First submitted 2008-09-28; First posted 2008-09-30 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Stroke, Acute; Infarction, Middle Cerebral Artery
MeSH Terms: conditions — Stroke; Infarction, Middle Cerebral Artery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- bone marrow stem cells (Other): Procedure: Infusion of autologous CD34+ stem cells into middle cerebral artery.
  Interventions: Procedure: Infusion on autologous CD34+ stem cells into middle cerebral artery

INTERVENTIONS:
Procedure: Infusion on autologous CD34+ stem cells into middle cerebral artery — Intraarterial infusion of autologous bone marrow stem cells into middle cerebral artery of acute stroke patients

SUMMARY:
The aim of the study is to determine the safety and efficacy on an autologous CD34+ subset bone marrow stem cell infusion into the middle cerebral artery in patients who have suffered acute middle cerebral artery stroke.

DETAILED DESCRIPTION:
The proposed trial will involve the recruitment of a total of 20 patients.

The cells will be collected from ten subject recruited as cases, via bone marrow sampling. The aspirate will be centrifuged on a Ficoll density gradient to isolate mononuclear cells, which will be resuspended in heparinized isotonic saline for infusion into the area of the stroke intra-arterially using the middle cerebral artery.

The investigators will monitor each case and control for a period of 6 months post-stem cell infusion. Initially, they will be subjected to a review after one month,three months and finally 6 months.

Assessment of adverse events will be by physical examination and measurement of laboratory parameters. Assessment of efficacy will be by physical examination and the measurement of laboratory, CT and MRI parameters.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and signs of clinically definite middle cerebral artery acute stroke.
* Time of stroke onset is known and treatment can be started between day 5 and 9 of onset.
* DWI-MRI has reliably shown relevant acute ischemic lesions
* Extracranial duplex/transcranial Doppler must confirm intra/extracranial arteries permeability.
* The stroke is severe (NIH Stroke Scale >= 8 before procedure).
* An age range of 18-80 years old.

Exclusion Criteria:

* Patients out of inclusion age range.
* Lacunar infarction.
* Patients with cancer.
* Patients with present or previous malignant disease during the last 5 years, except for basal cell carcinoma.
* Hematological causes of stroke.
* Severe co-morbidity.
* Hepatic or renal dysfunction.
* The patient is female and of childbearing potential (unless it is certain that pregnancy is not possible) or breast feeding.
* Patient is likely to be unavailable for follow-up.
* Patient with evidence of life threatening infection of life threatening illness.
* Patient was already dependent in activities of daily living before the present acute stroke.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Absence of new neurological deficits and adverse effects during the timeframe. | Duration of study

SECONDARY OUTCOMES:
Improvement in clinical function as assessed by the Modified Rankin Score, Barthel Scale and NIH stroke scale. | Duration of study

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospitales Universitarios Virgen del Rocío, Seville, Andalusia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias

REFERENCES:
- [Derived] Moniche F, Gonzalez A, Gonzalez-Marcos JR, Carmona M, Pinero P, Espigado I, Garcia-Solis D, Cayuela A, Montaner J, Boada C, Rosell A, Jimenez MD, Mayol A, Gil-Peralta A. Intra-arterial bone marrow mononuclear cells in ischemic stroke: a pilot clinical trial. Stroke. 2012 Aug;43(8):2242-4. doi: 10.1161/STROKEAHA.112.659409. Epub 2012 Jul 3. PMID 22764211
- [Derived] Mackie AR, Losordo DW. CD34-positive stem cells: in the treatment of heart and vascular disease in human beings. Tex Heart Inst J. 2011;38(5):474-85. PMID 22163120